CLINICAL TRIAL: NCT06174012
Title: The Effect of Sodium Fluoride Application on the Prevention of Radiation Caries in Nasopharyngeal Carcinoma Patients: A Prospective, Open, Randomized Controlled Phase II Trial
Brief Title: The Effect of Sodium Fluoride Application on the Prevention of Radiation Caries in NPC Patients
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Hai-Qiang Mai,MD,PhD, Professor, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2023-FXY-139
Record Dates: First submitted 2023-12-08; First posted 2023-12-18 (Actual); Last update posted 2023-12-18 (Actual); Status verified 2023-12

CONDITIONS: Sodium Fluoride
Keywords: Nasopharyngeal Carcinoma; Sodium Fluoride; Radiation Caries
MeSH Terms: conditions — Nasopharyngeal Carcinoma | interventions — Sodium Fluoride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sodium Fluoride Group (Experimental)
  Interventions: Drug: Sodium Fluoride
- Conventional care group (No Intervention)

INTERVENTIONS:
Drug: Sodium Fluoride — Sodium fluoride was applied before radiotherapy, at 3 months, 6 months, and 12 months after radiotherapy.
  Arms: Sodium Fluoride Group

SUMMARY:
To evaluate the efficacy of sodium fluoride to preventing radiation caries for patients with nasopharyngeal carcinoma receiving radiotherapy.

ELIGIBILITY:
Inclusion Criteria:

* a. Patients with histologically confirmed non-keratinizing NPC (including differentiated type and undifferentiated type, world health organization [WHO] II or III).

  b. Original clinical staged as II-IVa (according to the 8th AJCC edition) c. Male or female who are not pregnant. d. No evidence of distant metastasis (M0). e. Age between 18-60 years. f. WBC≥4×109/L, PLT≥100×109/L, HGB≥90g/L. g. Normal liver function test: Alanine Aminotransferase (ALT), Aspartate Aminotransferase (AST) <1.5×upper limit of normal (ULN) concomitant with alkaline phosphatase (ALP) ≤2.5×ULN, and bilirubin ≤ULN.

  i. With normal renal function test (creatinine clearance rate≥60 ml/min or creatinine< 1.5×ULN.

  j. The Eastern Cooperative Oncology Group (ECOG) Performance status less or equal to 1.

  k. Patients must be informed of the investigational nature of this study and give written informed consent.

  l. Patients receive nasopharyngeal and neck radiotherapy. m. After pre-radiotherapy oral examination, no less than 2 functional teeth in any 1/6 segment of the mouth.

Exclusion Criteria:

* a. With clinical stage of I and IVb (according to the 8 th AJCC edition). b. Patients with tumor recurrence or distant metastasis. c. Prior malignancy except adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer.

  d. History of previous radiotherapy (except for non-melanomatous skin cancers outside intended RT treatment volume).

  e. Prior chemotherapy or surgery (except diagnostic) to primary tumor or nodes. f. Pregnancy or lactation (consider pregnancy test in women of child-bearing age and emphasize effective contraception during the treatment period).

  g. Fewer than 2 functional teeth in any 1/6 segment of the mouth after pre-radiotherapy scaling.

  h. Lesions of infection in the oral cavity at baseline, severe gingivitis (gingival index = 3, i.e., severe inflammation of the gums, marked redness, swelling or ulceration of the gums, and a tendency to bleed automatically).

  i. Age < 18 or age > 60. j. Any severe intercurrent disease, which may bring unacceptable risk or affect the compliance of the trial, for example, unstable cardiac disease requiring treatment, acute exacerbation of chronic obstructive pulmonary disease or other respiratory illness requiring admission to hospital, renal disease, chronic hepatitis, diabetes with poor control (fasting plasma glucose >1.5×ULN), and mental disturbance.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 135 (Estimated)
Dates: Start 2023-12-15 (Estimated); Primary Completion 2024-11-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of radiation caries | 3、6、12 months after radiotherapy
  Incidence of radiation caries will be assessed by DMFT index.

SECONDARY OUTCOMES:
Correlation between radiation-induced otitis media and life quality after radiotherapy | 3、6、12 months after radiotherapy
  The life quality will be assessed by OHIP-14.

IPD SHARING:
Plan to Share IPD: No